CLINICAL TRIAL: NCT05657041
Title: Body Weight Adjusted Clopidogrel Treatment in Patients With Coronary Artery Disease
Acronym: BW-ACCORD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Collaborators: St. Antonius hospital Onderzoeksfonds (Unknown); Ace pharmaceuticals (Unknown); Allgen pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, Prof. dr., St. Antonius Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81095.100.22
Record Dates: First submitted 2022-11-18; First posted 2022-12-20 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease; Platelet Reactivity
Keywords: Antithrombotic Drugs; Pharmacodynamics; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: prospective, experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: body weight <60kg (Experimental): Treatment with clopidogrel 50mg once daily for a minimum of 10 days (max. 14 days), followed by a minimum of 10 days treatment with clopidogrel 25mg once daily (max 14 days).
  Interventions: Drug: Clopidogrel
- Group 2: body weight 60-100kg (No Intervention): Treatment with clopidogrel 75mg once daily
- Group 3: body weight >100kg (Experimental): Treatment with clopidogrel 150mg once daily for a minimum of 10 days (max. 14 days), followed by a minimum of 10 days treatment with prasugrel 10mg once daily (max 14 days).
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Body weight adjusted clopidogrel dosing
  Other Names: Prasugrel; Body weight adjusted
  Arms: Group 1: body weight <60kg; Group 3: body weight >100kg

SUMMARY:
Extreme body weights (BW) or body mass index (BMI) affect the pharmacokinetics of antithrombotic drugs and consequently may affect cardiovascular risk during treatment. The goal of this clinical trial is to establish if clopidogrel treatment can be optimized in patients with a low or high BW compared to patients with a normal BW by adjusting the dosage of clopidogrel and evaluating platelet reactivity.

Participants are stratified into three groups based on their BW (Low BW: BW <60kg; normal BW: 60-100kg; High BW: >100 kg)

Clopidogrel dosage will then be adjusted to the BW, as follows:

* Low BW: >10 days clopidogrel 50mg 1dd1, followed by >10 days clopidogrel 25mg 1dd1.
* Normal BW: Clopidogrel 75mg 1dd1.
* High BW: >10 days clopidogrel 150mg 1dd1 followed by >10 days prasugrel 10mg 1dd1.

The primary endpoint of the study is P2Y12 Reaction Units (PRU) and platelet inhibition measured using the VerifyNow measured before starting new treatment regimen (at the end of 10 days of treatment).

DETAILED DESCRIPTION:
Patients with a high BMI/BW have a higher cardiovascular risk and patients with a low BMI/BW seem to have a higher bleeding risk. A high BMI/BW affects the efficacy of clopidogrel. It is not yet known if this clopidogrel efficacy is altered in patients with a low BMI/BW and whether BW-adjusted treatment can optimise this efficacy. We hypothesize that a personalised treatment will eventually lead to a more optimal effect of clopidogrel, optimizing the balance between bleeding and thrombotic risk. This could benefit therapy compliance.

Primary Objective:

To determine if clopidogrel treatment can be optimized in patients with a low or high BW compared to patients with a normal BW by adjusting the dosage of clopidogrel and evaluating platelet reactivity measured using the VerifyNow.

Secondary Objective(s):

To determine if the CYP2C19 genotype has additional effect on the platelet reactivity in the different treatment groups.

This is a non-randomized single centre, prospective, experimental study in patients with CCS treated with clopidogrel 75mg (and aspirin). This study is designed to be pragmatic and is intended to be hypothesis generating. Patients have to be treated with clopidogrel for at least one month without the occurrence of a major bleeding event, an ischemic event (stroke, myocardial infarction, or coronary revascularization) and have to be free of angina complaints.

Participants are stratified into three groups based on their BW (Low BW: BW <60kg; normal BW: 60-100kg; High BW: >100 kg)

Clopidogrel dosage will then be adjusted to the BW, as follows:

* Low BW: >10 days clopidogrel 50mg 1dd1, followed by >10 days clopidogrel 25mg 1dd1.
* Normal BW: Clopidogrel 75mg 1dd1.
* High BW: >10 days clopidogrel 150mg 1dd1 followed by >10 days prasugrel 10mg 1dd1.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, ≥18 years of age
* Patients treated for CCS with clopidogrel 75mg QD (aspirin 100mg QD).
* Patients must be treated with clopidogrel 75mg for at least one month
* Patients must give consent by means of a signed informed consent

Exclusion Criteria:

* Contra-indication for aspirin
* Contra-indication for clopidogrel or prasugrel
* Occurrence of an ischemic event after PCI or ACS (stroke, myocardial infarction, or coronary revascularization)
* Presence of unstable angina complaints.
* Presence of two CYP2C19 Loss-of-function (LOF) alleles (*2 or *3)
* Scheduled for cardiac valve surgery
* Indication for chronic oral anticoagulants
* Expected life span of less than one year
* Pregnancy
* Suboptimal stent placement as determined by the cardiologist.
* Patients at increased risk of bleeding with two of the following characteristics: liver cirrhosis with portal hypertension, enhanced bleeding tendency, active malignancy in the past 12 months, thrombocytopenia, major surgery in the past month, spontaneous intracerebral haemorrhage, traumatic intracerebral haemorrhage in the past 12 months, major bleeding requiring hospitalisation or blood transfusion in the past month, ischaemic CVA in the past 5 months.
* Known with established stent thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | Baseline and 10 days after dose alteration
  Change in P2Y12 Reaction Units (PRU) measured using the VerifyNow
High on-treatment platelet reactivity (HTPR) | Baseline
  Number of participants with high on-treatment platelet reactivity (HTPR) defined by a PRU >208
High on-treatment platelet reactivity (HTPR) | 10 days
  Number of participants with high on-treatment platelet reactivity (HTPR) defined by a PRU >208
High on-treatment platelet reactivity (HTPR) | 20 days
  umber of participants with high on-treatment platelet reactivity (HTPR) defined by a PRU >208

SECONDARY OUTCOMES:
Bleeding complications | 30 days
  Number of participants with major or clinically relevant bleeding complications according to the Bleeding Academic Research Consortium Definition for Bleeding (BARC) classification.
Myocardial infarction | 30 days
  Number of participants with myocardial infarction as defined by the 4th Universal Definition of Myocardial Infarction
Stroke | 30 days
  Number of participants with stroke as defined by VARC definitions
Stent thrombosis | 30 days
  Number of participants with stent thrombosis as defined by ARC
All-cause death | 30 days
  Number of participants with all-cause death as defined by ARC

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - StAntoniusH, Nieuwegein, Utrecht
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No